CLINICAL TRIAL: NCT05261997
Title: Effect of Endotherapy on the Progression of Chronic Pancreatitis in Painless Patients
Brief Title: Endotherapy for Painless Chronic Pancreatitis
Acronym: EACH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Clinical Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Painless CP
Record Dates: First submitted 2021-11-24; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Pancreatitis, Chronic; Exocrine Pancreatic Insufficiency; Abdominal Pain; Cholangiopancreatography, Endoscopic Retrograde
Keywords: chronic pancreatitis; endoscopic retrograde cholangiopancreatography; Exocrine Pancreatic Insufficiency; painless
MeSH Terms: conditions — Pancreatitis, Chronic; Exocrine Pancreatic Insufficiency; Abdominal Pain | interventions — Lithotripsy; Cholangiopancreatography, Endoscopic Retrograde; Metformin

STUDY DESIGN:
Intervention Model Description: Patients will be divided into conservative treatment group or endoscopic treatment group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic group (Experimental): The patients received intravenous analgesia (flurbiprofen and remifentanil) before the ESWL (Compact Delta II; Dornier Med Tech, Wessling, Germany). After the last ESWL session, the patients are treated with following ERCP within 48h. ERCP was performed under conscious sedation with intramuscular administration of diazepam 2.5-5.0 mg and pethidine 25-50 mg. If necessary, endoscopic sphincterotomy was performed. A dilating bougie or balloon will be used to dilate the stenosis after sphincterotomy. Standard techniques (i.e., extraction basket, extraction balloon, or both) will be used for stone removal. A pancreatic duct stent for drainage and nasopancreatic catheters will be inserted for temporary drainage if necessary. Conservative treatments similar to patients in the control group were given in endoscopic group according to patients' condition.
  Interventions: Procedure: extracorporeal shock wave lithotripsy and endoscopic drainage of the main pancreatic duct
- Conservative group (Other): Patients will have pancreatic enzymes (Pancreatin Enteric-coated Capsules or Oryz-Aspergillus Enzyme and Pancreatin Table) to control symptoms of exocrine pancreatic insufficiency. The recommended initial dose for adults is (25 000-40 000) IU lipase per meal (40 000 IU for meals and 20 000 IU for snacks), which can be increased until the PEI is relieved. The maximum recommended dose is (75 000-80 000) IU lipase per meal. Actions including drugs(Acarbose Tablets, Glucophage, Glimepirde Tablets) or insulin(Biosynthetic Human Insulin Injection, Tresiba or both) would also be taken for control of diabetes according to patients' glucose levels.
  Interventions: Drug: pancreatic enzyme(Pancreatin Enteric-coated Capsules or Oryz-Aspergillus Enzyme and Pancreatin Table), antidiabetic medicine(Acarbose Tablets, Glucophage, Glimepirde Tablets)

INTERVENTIONS:
Procedure: extracorporeal shock wave lithotripsy and endoscopic drainage of the main pancreatic duct — In addition to drug administrated in the control group, patients in this group would be treated with ESWL and endoscopic drainage of the main pancreatic duct.
  Other Names: ESWL; ERCP
  Arms: Endoscopic group
Drug: pancreatic enzyme(Pancreatin Enteric-coated Capsules or Oryz-Aspergillus Enzyme and Pancreatin Table), antidiabetic medicine(Acarbose Tablets, Glucophage, Glimepirde Tablets) — Patients will receive drugs to control pancreatic insufficiency
  Arms: Conservative group

SUMMARY:
This is a prospective randomized controlled trial. . Patients will be divided into conservative or endoscopic group and fecal pancreatic elastase-1 (FE-1) is tested to evaluate pancreatic exocrine function. The effect of extracorporeal shock wave lithotripsy and endoscopic treatment on the progression of chronic pancreatitis in painless patients will be determined.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled trial. Patients will be divided into conservative or endoscopic group and FE-1 is tested to evaluate pancreatic exocrine function. The effect of extracorporeal shock wave lithotripsy and endoscopic treatment on the progression of chronic pancreatitis in painless patients will be determined.

Chronic pancreatitis (CP) is a pathologic fibro-inflammatory syndrome of the pancreas that eventually leads to damage of the gland in individuals with genetic, environmental and/or other risk factors. If widespread, this damage causes failure of exocrine and endocrine pancreatic function resulting in steatorrhea and diabetes. The global pooled incidence of CP is 10 cases [95% Confidence interval (CI) 8-12] per 100,000 general population per year. Endoscopic retrograde cholangiopancreatography (ERCP) and extracorporeal shock wave lithotripsy (ESWL) has become first-line therapy for patients with chronic pancreatitis according to guidelines. Endoscopic therapy has been proved effective and safe. The clearance rate of pancreatic stones was 42-76%, and the pain relief rate was 15-85%.

Pain is the major clinical features of CP and remained a major clinical challenge. It is present in up to 90% of patients and is the main cause of hospitalization in most patients.Patten of pain for patients with chronic pancreatitis differs widely.

However, some CP patients have never had abdominal pain during the course of the disease, and participants are often diagnosed with CP due to diabetes or steatorrhea, which are called painless CP, accounting for about 10% of the CP population. These patients are mainly characterized as pancreatic endocrine and exocrine insufficiency. Some studies proposed that painless CP may be related to the severity of inflammation and the pain sensitivity of patients, but the mechanism has not yet been elucidated.

It is still controversial whether painless CP requires active endoscopic intervention or not. The United European Gastroenterology evidence-based guidelines does not recommend endoscopic treatment in painless CP patients, but the recommendation is not supported by strong clinical research evidence. European Society of Gastrointestinal Endoscopy (ESGE) Guideline proposed whether active endoscopic treatment had a protective effect on the pancreatic function of patients with painless CP is still unconfirmed. On the contrary, a small sample study consisting of 41 CP patients by Katsushi found that endoscopic treatment can delay the progression of exocrine dysfunction in CP patients.Considering these contradicting results, it is urgent to conduct a clinical study to determine the effect of endoscopic treatment on preservation of pancreatic function in patients with CP.

Therefore, this study intends to use clinical prospective trials to explore whether patients with painless CP can benefit from active endoscopic minimally invasive interventions (including ERCP, ESWL, etc.), including slowing down the deterioration of pancreatic endocrine and exocrine function and improving patients' life quality and other aspects, and then provide an important reference basis for the clinical treatment of this type of patients.

Considering all these backgrounds, the primary outcome aimed to explore whether painless CP patients can benefit from endoscopic interventions (including ERCP, ESWL, etc.), including slowing down the deterioration of pancreatic endocrine and exocrine function, improving patients' life quality and other aspects. Based on the above, this study intends to provide important reference for the clinical treatment of painless CP patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with chronic pancreatitis without pain attack related with chronic pancreatitis;
* calcified stone in the cephalic or corporeal portion of the main pancreatic duct with upstream duct dilation;
* no ERCP or ESWL carried out before admission;

Exclusion Criteria:

* suspected to have malignant tumors;
* history of pancreatic surgery or gastrojejunostomy (Billroth II);
* with end-stage disease;
* pregnancy or lactation;
* refuse to write informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
exocrine function of the pancreas assessed by the value of fecal elastase in μg/g | 12 months
  Pancreatic exocrine function insufficiency(PEI) is defined as fecal elastase <200 μg/g. The result wii be divided into 4 conditions, including normal exocrine function, newly developed PEI, PEI relief, PEI persisting.

SECONDARY OUTCOMES:
endocrine function of the pancreas assessed by glycosylated hemoglobin in %. | 12 months
  It is considered as pancreatic endocrine function insufficiency when glycosylated hemoglobin >6.5%， the result of pancreatic endocrine function can also be divided into 4 parts similar to that of pancreatic exocrine function.
endocrine function of the pancreas assessed by fasting blood glucose in mmol/L | 12 months
  It is considered as pancreatic endocrine function insufficiency when fasting blood glucose >6.1mmol/L, the result of pancreatic endocrine function can also be divided into 4 parts similar to that of pancreatic exocrine function.
endocrine function of the pancreas assessed by fasting C peptide in ug/L | 12 months
  It is considered as pancreatic endocrine function insufficiency when fasting C peptide<1.1ug/L, the result of pancreatic endocrine function can also be divided into 4 parts similar to that of pancreatic exocrine function.
life quality assessed by SF-36 questionnaire | 12 months
  life quality assessed by the MOS item short from health survey (SF-36) questionnaire

OTHER OUTCOMES:
BMI in kg/m^2 | 12 months
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters.
Treatment-related costs in RMB from initial enrollment to the end of the study | 12 months
  The total costs in RMB of each hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, MD, Principal Investigator — Shanghai Changhai Hospital, Shanghai, China
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No